CLINICAL TRIAL: NCT03999476
Title: Randomized- Single Blind Trial of Ambu Ascope and Fiberoptic in Severely Difficult Air Way Patient Having Posterior Third Fixed Tongue Cancer
Brief Title: Evaluation of the Efficacy of Ambu® aScope for Intubation in Cancer Tongue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: mahmoud salem soliman (Other)
Collaborators: Cairo University (Other)
Responsible Party: Sponsor-Investigator, mahmoud salem soliman, Head of intensive care unit at new kaser al ainy teaching hospital , lecterur of anaesthesia and intensive care cairo universty ., Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: intubation in cancer tongue
Record Dates: First submitted 2019-06-22; First posted 2019-06-26 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Difficult Intubation

STUDY DESIGN:
Intervention Model Description: parallel assignment
Who Masked: Participant
Masking Description: patient will be under general anesthesia
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ambu scope (Experimental): intubation of cancer tongue patients with ambu scope device
  Interventions: Device: ambu ascope
- fiberoptic (Active Comparator): intubation of cancer tongue patients with fiberoptic device
  Interventions: Device: fibreroptic bronchoscope

INTERVENTIONS:
Device: ambu ascope — nasal route intubation by the device in fixed cancer tongue patients
  Other Names: Ambu® aScope™
  Arms: ambu scope
Device: fibreroptic bronchoscope — nasal route intubation by the device in fixed cancer tongue patients
  Arms: fiberoptic

SUMMARY:
This study compares the ascope with standard fiberscope using the nasal route of intubation in patient having sever difficult airway (having posterior one third cancer tongue with fixed mobility)

DETAILED DESCRIPTION:
patient will be allocated into two group according to the type of endoscope used group (F) fibro scope group and group (A) the ambu ascope group The timer will be started (T0), when touching the fiberscope or a scope. The standard fiberscope or a scope2 will be introduced through the nostril and advanced through the vocal cords, once carina identified the time will be recorded ( T1) When correct positioning of the trachea confirmed by detection of the end-tidal co2 curve on capnography (T2).

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients of ASA physical status I and II who will be scheduled for posterior third fixed cancer tongue with severe difficult airway requiring naso-tracheal intubation
2. aged 18-70 years

Exclusion Criteria:

1. ASA 2 or 4
2. pregnant

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2020-05-05 (Actual); Study Completion 2020-05-19 (Actual)

PRIMARY OUTCOMES:
time of successful intubation | 5 minutes
  measuring time in seconds for reaching carina and time for successful intubation
  .

SECONDARY OUTCOMES:
quality of vision | 5 minutes
  subjective assessment by operator
incidence of complications | 15 minutes
  accounting number of desaturation , bleeding , hypoxia .
easiness of intubation | 5 minutes
  subjective assessment
number of intubation trials | 30 minutes
  counting number of intubation in each group

CONTACTS AND LOCATIONS:
Overall Officials: Ekramy M Abdelghafar, MD, Principal Investigator — Cairo University
Locations (1):
- Kasr Alini Univeristy Hospital, Cairo, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data for primary and secondary outcome measures will be made available
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 3 months
Access Criteria: open

REFERENCES:
- [Background] Reeves DS, Brown NM. Mycobacterial contamination of fibreoptic bronchoscopes. J Hosp Infect. 1995 Jun;30 Suppl:531-6. doi: 10.1016/0195-6701(95)90059-4. PMID 7560994
- [Background] Han DW, Shim YH, Shin CS, Lee YW, Lee JS, Ahn SW. Estimation of the length of the nares-vocal cord. Anesth Analg. 2005 May;100(5):1533-1535. doi: 10.1213/01.ANE.0000149900.68354.33. PMID 15845720
- [Background] Marfin AG, Iqbal R, Mihm F, Popat MT, Scott SH, Pandit JJ. Determination of the site of tracheal tube impingement during nasotracheal fibreoptic intubation. Anaesthesia. 2006 Jul;61(7):646-50. doi: 10.1111/j.1365-2044.2006.04652.x. PMID 16792609